CLINICAL TRIAL: NCT01638143
Title: Comparison of Bioavailability of Three Different Vitamin K2 Formulations
Brief Title: Bio-equivalence Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 10-3-017
Record Dates: First submitted 2012-07-09; First posted 2012-07-11 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-07

CONDITIONS: Bioequivalence; Bioavailability
Keywords: vitamin K2; menaquinone-7; bioavailability

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Gnosis P-1000 capsules (Active Comparator): MK-7 capsules containing 75 µg of MK-7 (source: Gnosis, Italy).
  Interventions: Dietary Supplement: Gnosis P-1000 capsules
- Gnosis M1500 capsules (Active Comparator): MK-7 capsules containing 75 µg of MK-7 (source Gnosis, Italy).
  Interventions: Dietary Supplement: Gnosis M-1500 capsules
- MenaQ7 M-1500 capsules (Active Comparator): MK-7 capsules containing 75 µg of MK-7 (source: Nattopharma, Norway)
  Interventions: Dietary Supplement: MenaQ7 M-1500 capsules; Dietary Supplement: Gnosis P-1000 capsules

INTERVENTIONS:
Dietary Supplement: MenaQ7 M-1500 capsules — The study participants will receive three different types of capsules as a single dose (75 μg of MK-7/day):
  * MenaQ7 M-1500 capsule
  * Gnosis P-1000 capsule
  * Gnosis M-1500 capsule
  Every two weeks, participants switch to another type of capsule; the washout period will therefore be two weeks.
  Arms: MenaQ7 M-1500 capsules
Dietary Supplement: Gnosis P-1000 capsules — The study participants will receive three different types of capsules as a single dose (75 μg of MK-7/day):
  * MenaQ7 M-1500 capsule
  * Gnosis P-1000 capsule
  * Gnosis M-1500 capsule Every two weeks, participants switch to another type of capsule; the washout period will therefore be two weeks.
  Arms: Gnosis P-1000 capsules; MenaQ7 M-1500 capsules
Dietary Supplement: Gnosis M-1500 capsules — The study participants will receive three different types of capsules as a single dose (75 μg of MK-7/day):
  * MenaQ7 M-1500 capsule
  * Gnosis P-1000 capsule
  * Gnosis M-1500 capsule
  Every two weeks, participants switch to another type of capsule; the washout period will therefore be two weeks.
  Arms: Gnosis M1500 capsules

SUMMARY:
The primary objective of this study is to compare absorption of vitamin K2 (menaquinone-7) after intake of three different vitamin K2 supplements.

DETAILED DESCRIPTION:
Several manufacturers are producing vitamin K2 raw material in different forms, namely oil and powder. To ensure bioequivalence of different vitamin K2 sources, the investigators are interested to compare the bioavailability of three different vitamin K2 formulations that are already commercially available. Two different oils and one powder product will be compared in this randomized cross-over trial. The investigators hypothesize that different vitamin K2 sources give no differences in bioavailability of vitamin K2.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women, aged between 20 and 40 years
* Normal body weight and height (18.5 kg/m2 < BMI < 30 kg/m2)
* Stable body weight (weight gain or loss < 3 kg in past 3 mo)
* Written consent to take part in the study
* Agreement to adhere to dietary restrictions required by the protocol

Exclusion Criteria:

* Abuse of drugs and/or alcohol
* Use of vitamin supplements containing vitamin K
* Soy allergy
* Pregnancy
* a history of) metabolic or gastrointestinal diseases including hepatic disorders
* Chronic degenerative and/or inflammatory diseases, e.g. diabetes mellitus, renal failure
* Use of oral anticoagulants
* Corticoid treatment
* Subjects with anaemia or subjects who recently donated blood or plasma
* Systemic treatment or topical treatment likely to interfere with coagulation metabolism (salicylates, antibiotics)

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-11; Primary Completion 2011-01 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
MK-7 absorption profiles | 9 weeks
  The purpose of this study is to compare the MK-7 absorption profiles after intake of three different vitamin K2 (MK-7) products that are already on the market. The main study parameter is therefore the calculated AUC value from the individual MK-7 absorption profiles.

CONTACTS AND LOCATIONS:
Overall Officials: Cees Vermeer, PhD, Principal Investigator — VitaK BV Maastricht University
Locations (1):
- VitaK BV / Maastricht University Medical Center, Maastricht, Netherlands